CLINICAL TRIAL: NCT02102178
Title: Occupational Therapy Modulates the Pain in Cancer Patient Under Palliative
Brief Title: Occupational Therapy Modulates the Pain in Cancer Patient Under Palliative Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7683857344959085
Record Dates: First submitted 2014-03-27; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Cancer; Terminal Disease; Pain
Keywords: oncological pain; therapeutic activities; occupational therapy.
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Intensive occupational therapy) (Experimental): All patients received pharmacological treatment for pain in accordance with the World Health Organization (WHO)'s analgesic ladder and occupational therapy follow-up, with guidance regarding activities of daily living (ADLs).
  They also carried out therapeutic activities such as embroidery onto gauze (tapestry), weaving a scarf on a nail frame and playing dominos.
  Interventions: Other: Tapestry; Other: Regular occupation therapy; Other: Weaving a scarf on a nail frame; Other: Domino game
- Group 2 (Regular occupation therapy) (Active Comparator): All patients received pharmacological treatment for pain in according to WHO's analgesic ladder and only guidance regarding ADLs from the occupational therapist.
  Interventions: Other: Regular occupation therapy

INTERVENTIONS:
Other: Tapestry — A gauze screen, wool thread appropriate for tapestry and a large needle were used.
  The entire screen was filled with a striped pattern made of embroidered half-stitches in the individuals' preferred colors. To fill the screen with half-stitches, the needle was always worked in diagonal movements, point to point. The stitches were started keeping a distance of three points from the four edges.
  Arms: Group 1 (Intensive occupational therapy)
Other: Regular occupation therapy — All the patients were followed up daily for 10 days by a single occupational therapist for around 30 minutes, during which they received guidance regarding how best to perform their ADLs, i.e. how to position themselves when sitting down and standing up, dressing and undressing, feeding themselves, performing personal hygiene and undertaking leisure activities, with the aim of protecting their joints, reducing the pain and expending less energy.
  Other Names: Occupational therapy
Other: Weaving a scarf on a nail frame — Weaving a scarf on a nail frame: this activity used a rectangular wooden frame (30 cm x 10 cm), with an empty space in the middle and nails distributed at 1 cm intervals along all sides, together with a crochet needle and wool thread.
  Procedure: The thread was measured out on the frame and all the fringes were cut to the same length. After this, each thread was knotted, leaving a loop that was placed over each nail. A wool thread was tied to the nail at the corner and a zigzag pattern was woven between alternate nails. On the return, the zigzag weave went via the nails that had initially been missed out. Using the crochet needle, the loop of the fringe was pulled across on top of the zigzag. The scarf went on coming out from under the frame. The zigzag sequence and the needle movement were repeated until the scarf reached the desired length.
  Arms: Group 1 (Intensive occupational therapy)
Other: Domino game — Each player received seven dominos and kept them concealed from the adversaries' eyes. The player with the double-six (domino with the number six at both ends) started the game. If this domino had not been dealt out to any player, the one with the highest double domino started. Following on from this first player, in clockwise direction, each subsequent player placed one domino at one of the ends of the chain that was formed as the dominos were played. If a player did not have a domino that could be played, he would go to the pile and keep on picking up dominos until getting one that would fit. If no such domino existed, the player would then pass his turn on to the next player. The first player to get rid of all his dominos was the winner. If the game became "blocked", i.e. there was no longer any possibility of adding dominos to the chain, the points in each player's hand were counted and the winner was the one with the lowest number of points in his hand.
  Arms: Group 1 (Intensive occupational therapy)

SUMMARY:
Pain is one of the most incapacitating symptoms because it is a complex experience that includes sensory and emotional perceptions, in which sensory, affective, cognitive, behavioral, cultural and social characteristics interact. Around 79% of advanced cancer cases present pain.

There is evidence that non-pharmacological therapeutic activities are useful for controlling oncological pain and other symptoms resulting from such diseases.

This study evaluated the results relating to pain modulation and improvement of emotional symptoms and quality of life, from an occupational therapy program applied to oncological patients who were receiving palliative care.

DETAILED DESCRIPTION:
Occupational therapy provides a variety of practical and psychosocial interventions to enable individuals to adapt to the difficulties that result from advanced disease. In this form of therapy, the use of certain manual play activities are highlighted as a working tool, with the aim of intervening in relation to the limitations and/or physical and psychological diseases. Such interventions may transform some of these patients' interests in life, facilitate the development of undiscovered talents and skills and allow them to discover their artistic, artisanal or physical potentials.

The role and interventions of occupational therapy within palliative care are wide-ranging and challenging, with a vocation to help individuals to value the remainder of their lives and live for the present moment in the best way possible, through providing options for them to keep themselves in a physical and emotional condition that allows them to carry out activities that would be gratifying and stimulating. The effects from this will assist them in preparing for the end of life with more dignity and respect.

The relevance of occupational therapy interventions in relation to oncology and, in particular, palliative care has been little studied. However, it is known that this may contribute towards improving the quality of life in interpersonal relationships and diminishing pain and distress, through providing guidance regarding activities of daily living and through the use of therapeutic activities, especially in relation to hospitalization processes.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* advanced neoplasia without therapeutic possibilities for cure
* intensity of pain greater than or equal to 5 on the 10-centimeter VAS.
* expected to live for more than three months,
* Karnofsky Performance Status (KPS) of between 40 and 70%
* Patients not candidate to palliative and antalgic chemotherapy and/or radiotherapy.
* Patients or their legal representatives must be able to read, understand and provide written informed consent to participate in the study.

Exclusion Criteria:

* Presence of aphasia and/or severe visual disturbances;
* Patients admitted to hospital for pain control in situations considered to be pain emergencies such as bone fracture, infection, medullary compression or metastasis in the central nervous system
* Patients with poor cognitive capacity (unable to understand the research questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Before and after occupational therapy intervention every day up to day 10
  The pain intensity was assessed every day before and after each intervention by means of the 10 cm VAS. The McGill pain questionnaire was used on the first and last (tenth) day of the study.

SECONDARY OUTCOMES:
Quality of life score | Baseline and day 10
  Quality of life was evaluated by means of the SF-12 Health Survey, which is a shortened version of the SF-36 Health Survey.
Anxiety rate | Baseline and day 10
  The anxiety symptoms were assessed using the Hospital Anxiety and Depression Scale (HADS).
Depression rate | Baseline and day 10
  The depression symptoms were assessed using the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Takeda, Occupational Therapy, Principal Investigator — Barretos Cancer Hospital; Maria Salete A. Nascimento, PhD, Principal Investigator — Barretos Cancer Hospital

REFERENCES:
- [Background] Kasven-Gonzalez N, Souverain R, Miale S. Improving quality of life through rehabilitation in palliative care: case report. Palliat Support Care. 2010 Sep;8(3):359-69. doi: 10.1017/S1478951510000167. PMID 20875180
- [Background] Sviden GA, Tham K, Borell L. Involvement in everyday life for people with a life threatening illness. Palliat Support Care. 2010 Sep;8(3):345-52. doi: 10.1017/S1478951510000143. PMID 20875178
- [Background] Halkett GK, Ciccarelli M, Keesing S, Aoun S. Occupational therapy in palliative care: is it under-utilised in Western Australia? Aust Occup Ther J. 2010 Oct;57(5):301-9. doi: 10.1111/j.1440-1630.2009.00843.x. PMID 20868419
- [Background] Meredith PJ. Has undergraduate education prepared occupational therapy students for possible practice in palliative care? Aust Occup Ther J. 2010 Aug;57(4):224-32. doi: 10.1111/j.1440-1630.2009.00836.x. PMID 20854596
- [Background] Kumano K, Matsuda N, Matsumoto H, Noguchi A, Tada Y, Koezuka M, Sano K, Kasamatu Y. [The role of occupational therapist in Palliative Care Team]. Gan To Kagaku Ryoho. 2010 Sep;37(9):1825-7. No abstract available. Japanese. PMID 20841957
- [Background] Kuhara S, Kakou H, Tokuo M, Nogami M, Takemura J, Hachisuka K. [Palliative rehabilitation of two patients with terminal stage cancer: a visit to patient's home and the provision of advice by a nurse and rehabilitation staff members before discharge--from physical therapist's perspective]. J UOEH. 2009 Dec 1;31(4):359-64. doi: 10.7888/juoeh.31.359. Japanese. PMID 20000010